CLINICAL TRIAL: NCT05456165
Title: A Randomized, Open-Label, Phase 2 Study of a Patient-Specific Vaccine Targeting Neoantigens in Combination With Immune Checkpoint Blockade for Patients With Colon Cancer With Minimal Residual Disease Following Surgical Resection and Standard Adjuvant Chemotherapy
Brief Title: Study of an Individualized Vaccine Targeting Neoantigens in Combination With Immune Checkpoint Blockade for Patients With Colon Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: terminated due to reprioritization
Sponsor: Gritstone bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO-008; GRANITE-ADJUVANT (Other: Gritstone)
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Colonic Neoplasms; Colorectal Neoplasms
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms | interventions — atezolizumab; Ipilimumab; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GRT-C901/GRT-R902 Vaccine arm (Experimental): After surgical resection, patients who are circulating tumor DNA (ctDNA) positive will receive adjuvant chemotherapy for 12-24 weeks during which they will undergo neoantigen prediction, randomization, and vaccine manufacturing. After study treatment screening, patients who are still ctDNA positive with no evidence of residual or metastatic disease will receive a total of 6 doses of GRT-C901/ GRT-R902, 2 doses of ipilimumab, and 13 doses of atezolizumab. Study visits occur every 28 days.
  Interventions: Drug: GRT-C901; Drug: GRT-R902; Drug: Atezolizumab; Drug: Ipilimumab; Drug: Adjuvant chemotherapy
- Observation arm (Active Comparator): After surgical resection, patients who are ctDNA positive will receive adjuvant chemotherapy for 12-24 weeks during which they will undergo neoantigen prediction and randomization. After study treatment screening, patients who are still ctDNA positive with no evidence of residual or metastatic disease will be observed via study visits occur every 12 weeks.
  Interventions: Drug: Adjuvant chemotherapy

INTERVENTIONS:
Drug: GRT-C901 — An individualized neoantigen cancer vaccine using an adenovirus vector administered via intramuscular (IM) injections at Visit 1 and boost at Visit 6.
  Arms: GRT-C901/GRT-R902 Vaccine arm
Drug: GRT-R902 — An individualized neoantigen cancer vaccine using a self-amplifying mRNA (samRNA) vector administered via IM injection at Visits 2, 4, 9, and 12.
  Arms: GRT-C901/GRT-R902 Vaccine arm
Drug: Atezolizumab — Dose of 1680 mg administered once every 4 weeks (Q4W) via intravenous (IV) infusion at Visits 1-13.
  Arms: GRT-C901/GRT-R902 Vaccine arm
Drug: Ipilimumab — Dose of 30 mg administered via subcutaneous (SC) injection only with the first dose of GRT-C901 at Visit 1 and GRTR902 at Visit 2.
  Arms: GRT-C901/GRT-R902 Vaccine arm
Drug: Adjuvant chemotherapy — Administered according to standard of care.

SUMMARY:
The primary objective is to assess and characterize the antitumor activity and safety and tolerability of adjuvant treatment with an individualized neoantigen vaccine called GRT-C901/GRT-R902 (chimpanzee adenovirus [ChAd] and self-amplifying messenger RNA [samRNA] vectors), in combination with checkpoint inhibitors. Antitumor activity will be based on molecular response in patients with colon cancer who have circulating tumor deoxyribonucleic acid (ctDNA) following surgical resection.

DETAILED DESCRIPTION:
Tumors harboring non-synonymous deoxyribonucleic acid (DNA) mutations present peptides containing these mutations as non-self antigens in the context of human leukocyte antigens (HLAs) on the tumor cell surface. A fraction of mutated peptides results in neoantigens capable of generating T cell responses that exclusively target tumor cells. Sensitive detection of these mutations allows for the identification of neoantigens unique to each patient's tumor to be included in a personalized cancer vaccine that targets these neoantigens. This vaccine regimen uses two vaccine vectors as a heterologous prime/boost approach (GRT-C901, ChAd as prime and GRT-R902, samRNA as boost) to stimulate an immune response. This study (GRANITE-ADJUVANT) will explore the anti-tumor activity of this individualized, patient specific immunotherapy in combination with checkpoint inhibitors.

ELIGIBILITY:
Inclusion Criteria

For Vaccine Production Stage:

* Patients with a high-risk stage II or stage III colon cancer, including high-risk stage II colon cancer defined as meeting any of the following criteria: T4 tumors, Grade ≥3, clinical presentation with bowel obstruction or perforation, histological signs of vascular or lymphatic or perineural invasions, and <12 nodes examined
* Patient has evidence of minimal residual disease (MRD) prior to initiating adjuvant chemotherapy (ACT) based on the presence of ctDNA
* Patient has received approximately <6 weeks of ACT.
* Margin negative (R0) pathology on resection
* Availability of formalin fixed, paraffin embedded (FFPE) tumor specimens
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 or equivalent for patients 12 to 17 years of age
* Patient has adequate organ function as defined by: peripheral white blood cell (WBC) count ≥3000/mm^3, absolute lymphocyte count (ALC) ≥800/mm^3, absolute neutrophils count (ANC) ≥1500/mm^3, platelets ≥100,000/mm^3, hemoglobin ≥9 g/dL, albumin ≥3 g/dL, calculated creatinine clearance >50 mL/min using Cockcroft-Gault equation, alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤3 × upper limit of normal (ULN), total serum bilirubin ≤1.5 × ULN OR direct bilirubin ≤1 × ULN, international normalized ratio (INR), prothrombin time (PT), or partial thromboplastin time (PTT) ≤1.5 × ULN, unless patient is receiving anti-coagulant therapy, in which case patients are eligible if PT and PTT are within therapeutic range of intended use of anti-coagulants, and carcinoembryonic antigen levels ≤1.5 × ULN.
* A woman of childbearing potential (WCBP) must be willing to undergo pregnancy testing and agrees to the use at least 1 highly effective contraceptive method during the study treatment period and for 5 months after last investigational study treatment

For Study Treatment Stage:

* Have a confirmed diagnosis of high-risk stage II or stage III micro-satellite stable (MSS)-colon cancer and have had their tumor surgically resected, have completed standard ACT and have no evidence of disease radiographically, and have evidence of MRD based on detection of ctDNA following ACT
* ECOG performance status of 0 to 1 or equivalent for patients 12-17 years of age
* Have adequate organ function with peripheral WBC count ≥2000/mm^3, ALC ≥500/mm^3, ANC ≥1000/mm^3, platelets ≥75,000/mm^3, hemoglobin ≥9 g/dL, albumin ≥3 g/dL, calculated creatinine clearance >40 mL/min using Cockcroft-Gault equation, ALT and AST ≤3 × ULN, total serum bilirubin ≤1.5 × ULN OR direct bilirubin ≤1 × ULN, and INR, PT, or PTT ≤1.5 × ULN
* If a WCBP, must be willing to undergo pregnancy testing and agrees to the use at least 1 highly effective contraceptive method during the study treatment period and for 5 months after last investigational study treatment
* If male and sexually active with a WCBP, must agree to use highly effective contraception such as latex condom plus partner use of a highly effective contraceptive method during the study treatment period and for 5 months after last investigational study treatment.

Exclusion Criteria

For Vaccine Production Stage:

* Patients with micro-satellite instable (MSI)-high disease
* Patients with known tumor mutational burden (TMB) <1 non-synonymous mutations/megabase
* Patients with known DNA Polymerase Epsilon mutations
* Known exposure to chimpanzee adenovirus (ChAd) within the prior 6 months, plan to receive a ChAd-based vaccine in the next 6 months, and/or any history or anaphylaxis in reaction to a vaccination
* Bleeding disorder or history of significant bruising or bleeding following intramuscular (IM) injections or blood draws
* Immunosuppression anticipated at time of study treatment
* Patient has received prior therapy consisting of anti-cytotoxic T lymphocyte-associated antigen (CTLA-4), anti-programmed cell death-1 receptor (PD-1), anti-programmed death ligand-1(PD-L1), or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* History of allogeneic tissue/solid organ transplant
* Active or history of autoimmune disease or immune deficiency
* History of other cancer within 2 years
* Active tuberculosis or recent (<2 week) clinically significant infection, or evidence of active hepatitis B or hepatitis C or known history of positive test for human immunodeficiency virus (HIV) if CD4+ T-cell count is ≤200 cells/microliter.
* History of pneumonitis requiring systemic steroids for treatment (with the exception of prior resolved in-field radiation pneumonitis)
* Myocardial infarction within 3 months or prior to study treatment, unstable angina, serious uncontrolled cardiac arrhythmia, history of myocarditis, or congestive heart failure (New York Heart Association [NYHA] Grade 3 and 4)
* Pregnant, planning to become pregnant, or nursing

For Study Treatment Stage

* Patient is receiving treatment with investigational products and/or other anti-cancer therapies.
* Known exposure to ChAd within the prior 6 months, plan to receive a ChAd-based vaccine in the next 6 months, and/or any history or anaphylaxis in reaction to a vaccination
* Immunosuppression from concurrent, recent (≤4 weeks) or anticipated treatment with systemic corticosteroids or other immunosuppressive medications or conditions such as hypogammaglobulinemia, or radiation exposure
* Patients who have not recovered from prior cancer therapy-induced AEs
* Any severe concurrent non-cancer disease
* Active tuberculosis or recent (<2 weeks) clinically significant infection, evidence of active hepatitis B or hepatitis C, or known history of positive test for HIV if CD4+ T-cell count is ≤200 cells/microliter
* History of pneumonitis requiring systemic steroids for treatment
* Myocardial infarction within 6 months prior to initiating study treatment, unstable angina, serious uncontrolled cardiac arrhythmia, history of myocarditis, or congestive heart failure (NYHA Grade 3 and 4).
* Pregnant, planning to become pregnant, or nursing

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Patients with a ≥50% Decrease from Baseline in Circulating Tumor deoxyribonucleic acid (ctDNA) | Baseline and up to ~24 months
Incidence and Severity of Adverse Events | Up to ~100 days after last study treatment (Up to 62 weeks)
  The incidence and severity will be assessed for treatment-emergent adverse events (TEAEs), immune-related AEs (irAEs), treatment-related AEs, serious AEs (SAEs), AEs leading to death while patients are on treatment or up to 100 days after the last study treatment, AEs leading to dose delays or dose discontinuation, and AEs leading to discontinuation of study treatment using National Cancer Institute (NCI) Criteria for Adverse Events (CTCAE) v5.0

SECONDARY OUTCOMES:
Recurrence-free survival (RFS) per Investigator | From time of randomization until first recurrence of the same cancer, or death (Up to ~36 months)
Disease-free survival (DFS) per Investigator | From time of randomization until first recurrence of any cancer, or death (Up to ~36 months)
Overall Survival (OS) | From time of randomization until death due to any cause (Up to ~36 months)
Conversion of Patients with ctDNA at Baseline to Undetectable ctDNA as Assessed via a Polymerase Chain Reaction (PCR)-Based Assay | Baseline and up to ~24 months
Longest Duration of Molecular response of ctDNA Decrease from Baseline | Baseline and up to ~24 months
Success of Vaccine Manufacture | Up to 28 days before Day 1 of study drug administration
  Vaccine manufacture success measured by the number of patients having sufficient neoantigens identified to warrant vaccine production.
T-cell response using Peripheral Blood Mononuclear Cells (PBMCs) | Up to ~24 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - NYU Langone Health, New York, New York
  - Christ Hospital Cancer Center, Cincinnati, Ohio